CLINICAL TRIAL: NCT03535454
Title: Work-Related Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Fibromyalgia, Secondary
Keywords: Fibromyalgia; Musculoskeletal Diseases; Work
MeSH Terms: conditions — Fibromyalgia; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Factory workers
  Interventions: Other: working hours
- Nurses
  Interventions: Other: working hours
- Janitors
  Interventions: Other: working hours
- Data automation employees
  Interventions: Other: working hours

INTERVENTIONS:
Other: working hours — weekly working hours

SUMMARY:
The research is about fibromyalgia prevalency in working population and searching work-related fibromyalgia.

DETAILED DESCRIPTION:
4 different job population will be included in the study. Totally 200 people wil be included and evaluated. All participants will be women. The investigators will diagnose fibromyalgia with 2016 updated diagnostic criteria and evaluate work related musculoskeletal pain with nordic musculoskeletal questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* working at least 3 months in same working place

Exclusion Criteria:

* Diagnosed with the other musculoskeletal diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Working woman
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
work related fibromyalgia | 3 months
  fibromyalgia in working population

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No